CLINICAL TRIAL: NCT01080859
Title: Early Coverage and Vessel Wall Response of the Bio-Active-stent and Everolimus-Eluting Stent Implanted in Acute Coronary Syndrome Assessed By Optical Coherence Tomography (BASE-OCT)
Brief Title: Vessel Wall Response of the Bio-Active-stent and Everolimus-Eluting Stent Assessed By Optical Coherence Tomography
Acronym: BASE-OCT
Status: Completed | Type: Observational
Sponsor: The Hospital District of Satakunta (Other)
Responsible Party: Satakun Hospital District, Satakunta Central Hospital
Other Study IDs: SA-004
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Acute Coronary Syndrome
Keywords: titanium; everolimus; oct; acute coronary syndrome; stent; pci; stenting
MeSH Terms: conditions — Acute Coronary Syndrome; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- BAS: Patient's receiving BAS
  Interventions: Device: OCT
- EES: Patients receiving EES
  Interventions: Device: OCT

INTERVENTIONS:
Device: OCT — Optical coherence tomography
  Other Names: TITAN-2, Hexacath, France
  Groups: BAS
Device: OCT — Optical coherence tomography
  Other Names: Xience-V, Abbott vascular, USA
  Groups: EES

SUMMARY:
The purpose of the trial is to evaluate the completeness of struts coverage and vessel wall response (strut malapposition, neoin-timal formation) to the bio-active-stent (BAS) versus ever-olimus-eluting stent (EES) implanted for the treatment of the culprit lesion in acute coronary syndrome.

DETAILED DESCRIPTION:
A prospective, randomized and controlled study comparing the coverage of the BAS and EES implanted in acute coronary syndrome.

Clinical follow-up at 1, 6, 12 and 18 months. OCT analysis at the time of the 6 to 8 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old;
* The patient is presenting with acute coronary syndrome, and according to hospital routine practice, eligible for percutaneous coronary intervention;
* Patient or the patient's legal representative has been informed of the nature of the study and has provided written informed consent as approved by the Institutional Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Lesions in coronary artery bypass grafts
* Left main disease
* Killip class III-IV
* Allergy to aspirin / thienopyridine
* Patient in anticoagulation therapy
* No suitable anatomy for OCT scan
* Ostial lesion
* Tortuosity anatomy
* Very distal lesion
* Vessel size > 3.75 mm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with acute coronary syndrome and who were treated either BAS or EES during the index PCI.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Uncovered stent struts | 6-8 months
  OCT number of uncovered stent struts for BAS versus EES.

SECONDARY OUTCOMES:
Cardiac death,MI, stent thrombosis (ST) and TLR. | 1, 6, 12 and 18 months
  Device oriented composite endpoint, defined as cardiac death,MI, stent thrombosis (ST) and TLR at at 1, 6, 12 and 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pasi P Karjalainen, MD, PhD, Principal Investigator — Satakunta Central Hospital, Pori, Finland; Antti Ylitalo, MD, PhD, Study Chair — Satakunta Central Hospital, Pori, Finland
Locations (1):
- Satakunta Central Hospital, Pori, Finland

REFERENCES:
- [Derived] Karjalainen P, Kiviniemi TO, Lehtinen T, Nammas W, Ylitalo A, Saraste A, Mikkelsson J, Pietila M, Biancari F, Airaksinen JK. Neointimal coverage and vasodilator response to titanium-nitride-oxide-coated bioactive stents and everolimus-eluting stents in patients with acute coronary syndrome: insights from the BASE-ACS trial. Int J Cardiovasc Imaging. 2013 Dec;29(8):1693-703. doi: 10.1007/s10554-013-0285-8. Epub 2013 Aug 31. PMID 23996244